CLINICAL TRIAL: NCT00130715
Title: A Prospective, Randomized, Multicenter, Controlled Evaluation of the Efficacy and Safety of Seprafilm in the Reduction of Incidence of Bowel Obstruction in General Surgery
Brief Title: Seprafilm in the Reduction of Incidence of Bowel Obstruction in General Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SF97-0601
Record Dates: First submitted 2005-08-15; First posted 2005-08-16 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Intestinal Obstruction; Digestive System Surgical Procedures
Keywords: Patients undergoing a variety of abdominal surgical procedures
MeSH Terms: conditions — Intestinal Obstruction

INTERVENTIONS:
Device: Seprafilm Bioresorbable Membrane

SUMMARY:
The purpose of the study is to evaluate the efficacy of Seprafilm in reducing the incidence of bowel obstruction and to evaluate the incidence of all serious adverse events (SAEs) associated with the use of Seprafilm occurring within 30 days postoperatively, and the incidence of abdominopelvic abscess within 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were undergoing colon and/or rectal resections and/or adhesiolysis for treatment of bowel obstruction

Exclusion Criteria:

* Patients with any medical condition or disease where 5-year survival was not expected
* Patients undergoing laparoscopy
* Patients undergoing surgery for treatment of acute abdominal trauma
* Patients with an abscess (abdominal or pelvic) present during the initial surgery
* Patients with a history of pulmonary embolus or deep vein thrombosis (DVT) within 1 year of surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-06; Study Completion 2003-08

PRIMARY OUTCOMES:
Reducing the incidence of bowel obstruction following intestinal resection, and subsequently, reducing the number of re-operations

CONTACTS AND LOCATIONS:
Locations (21):
- United States (16):
  - Mayo Clinic, Scottsdale, Arizona
  - Kaiser Permanente Medical Center, Los Angeles, California
  - USC School of Medicine, Los Angeles, California
  - Harbor UCLA, Torrence, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Cleveland Clinic, Weston, Florida
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Medical Center, Rochester, Minnesota
  - Colon & Rectal Surgery Associates, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas Medical School, Houston, Texas
- Mount Sinai Hospital, Toronto, Ontario, Canada
- University of Erlangen, Erlangen, Germany
- University Hospital Nijmegen, Nijmegan, Netherlands
- United Kingdom (2):
  - University of Hull, Hull
  - St. Mary's Hospital, London